CLINICAL TRIAL: NCT01159587
Title: Observational Study Evaluating Efficacy and Costs of Secondary Prophylaxis vs On-demand Therapy With Kogenate Bayer in Patients With Severe Haemophilia A. POTTER
Brief Title: Prophylaxis Versus On-demand Therapy Through Economic Report
Acronym: POTTER
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayser Schering Pharma AG
Other Study IDs: 11856
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222)
- Group 2
  Interventions: Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Long-term secondary prophylaxis with product administered 20-30 UI /kg three times weekly
  Groups: Group 1
Drug: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — On-demand treatment with product given only for bleeding episodes
  Groups: Group 2

SUMMARY:
The project is a controlled observational, multicenter, prospective data collection on secondary prophylaxis with Kogenate Bayer in adolescents and adults with severe haemophilia A (FVIII < 1%).

The observational period will cover at least 5 years per patient.

The long-term secondary prophylaxis group will be compared versus on-demand treatment group by the assessment of orthopedic status progression and pharmacoeconomics evaluation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 12 years and ≤ 55 years
* severe haemophilia A (FVIII < 1%)
* absence of inhibitors (Bethesda titre < 0.6 BU/ml)
* Previous Treated Patients (prior exposure days > 200)
* Kogenate Bayer administered 20-30 IU/kg -3 times a week, for the prophylaxis group
* ≥ 6 joint bleeds requiring treatment with FVIII concentrates in the previous 6 months before enrollment, for on-demand group
* written informed consent

Exclusion Criteria:

* concomitant severe and chronic diseases or congenital skeletal malformation
* unreliability of patient or likelihood of follow-up failure
* presence of inhibitors or history of inhibitors (in the previous 2 years)
* currently on immune tolerance treatment
* hepatic cirrhosis or liver disease in rapid progression
* AIDS
* platelet count < 75,000/mm3
* presence of conditions that influence negatively patient´s compliance
* participation in another study

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Haemophilics
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2004-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy, safety and pharmacoeconomic of long-term secondary prophylaxis with Kogenate Bayer in comparison to on-demand treatment with Kogenate Bayer in terms of joint bleeding episodes per year | Every 6 months

SECONDARY OUTCOMES:
Efficacy, safety, pharmacoeconomic impact of secondary prophylaxis versus on demand group in terms of overall bleeding episodes | Every 6 months
Muscolo skeletal evaluation by Orthopedic Joint Score | Every 12 months
Radiological Evaluation by Pettersson Score | Baseline and after 3-5 years
Health related quality of life | Every 12 months
cost-effectiveness and utility, patient compliance, adverse events | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Italy

REFERENCES:
- [Derived] Tagliaferri A, Feola G, Molinari AC, Santoro C, Rivolta GF, Cultrera DB, Gagliano F, Zanon E, Mancuso ME, Valdre L, Mameli L, Amoresano S, Mathew P, Coppola A; POTTER Study Group. Benefits of prophylaxis versus on-demand treatment in adolescents and adults with severe haemophilia A: the POTTER study. Thromb Haemost. 2015 Jul;114(1):35-45. doi: 10.1160/TH14-05-0407. Epub 2015 Apr 9. PMID 25855376